CLINICAL TRIAL: NCT03524781
Title: Treatment of Newly Diagnosed Gastroesophageal Reflux Disease in a National Population-based Cohort
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Kolding Sygehus (Other); Odense Patient Data Explorative Network (Other)
Responsible Party: Principal Investigator, Jonas Sanberg Jensen, MD, PhD Student, University of Southern Denmark
Other Study IDs: JSJ_OP445
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Gastroesophageal Reflux
Keywords: Anti-reflux surgery; Proton-pump inhibitors; Upper endoscopy
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the treatment of newly diagnosed gastro-esophageal reflux disease in a Danish national cohort, comparing medical and surgical treatment.

DETAILED DESCRIPTION:
Aim: To compare rate of surgery with medical treatment in patients with newly diagnosed gastro-esophageal reflux disease in a nationwide population based cohort over 15 years.

Background: Between 1990 and 1997, frequency of anti-reflux surgery in USA rose from 4,4 per 100.000 inhabitants to 12 per 100.000 inhabitants. In the same period a trans-abdominal laparoscopic approach increased to 64% of cases and mortality as well as morbidity decreased. The operation rate peaked around 2000 with an increase of 260% to approximately 16.7 operations per 100.000 inhabitants. Complications fell to its lowest point around 2000 as well.

Hereafter, the frequency of anti-reflux surgery dropped by 40% between 2000 and 2006. Complications in the form of morbidity and mortality rates steadily rose again, but the patients having performed surgery were now older and have longer hospital stays and more comorbidity. A slight rise in frequency of anti-reflux surgery to 6,1 per 100.000 inhabitants was registered in 2010 and at this time length of stay, morbidity and mortality rates have decreased, probably illustrating an increased experience. Interesting to note is, that in the American data, use of laparoscopic approach does tend to plateau at 70-80%.

It is unknown whether anti-reflux surgery in Denmark has followed the same trend. There are important differences in the setup of surgical service that may affect the results, as open anti-reflux surgery never gained much popularity in Denmark. Also, significantly fewer centers offer the procedure. In a study of re-operative anti-reflux surgery based on data from 1997-2005, a primary anti-reflux surgery rate of 5.2 per 100.000 inhabitants was reported. However, we do not know how this rate has developed or was preceded.

Hypothesis: From 2000-2015 there has been an increase in diagnosis of GERD and in the use of anti-secretory drugs, but a decrease in the utilization of anti-reflux surgery.

Methods and materials: Patient selection will be done through the Danish National Patient Registers. Included will be the period 2000-2015 for a total of 15 years of follow-up.

All adult Danish patients diagnosed with GERD and GERD-related diagnosis will be identified (ICD-10 DK21.0-21.9B & DK20.9B) using The National Patient Registry.To validate GERD-diagnosis, upper endoscopy must have been performed no more than three months before time of diagnosis.

Patients with GERD-diagnosis within previous four years or with concomitant diagnosis requiring independent anti-secretory treatment will be excluded (DK25.0-9, DK26.0-9, DK27.0-9, DK22.7 & DE16.4B). Patients diagnosed with cancer of the gastrointestinal tract (DC15-26) will also be excluded.

Using the Danish National Prescription Register, use of H2-antagonists (A02BA), proton pump inhibitors (A02BC), prostaglandins A02BB and bismuth, alginate and sucralfate (A02BX) will be identified in daily doses within two years of GERD-diagnosis. Anti-reflux surgery within the same period will be identified from The National Patient Registry using the procedure codes (NOMESCO: KJBC00, KJBC01, KJBC02, KJBW96, KJBW97).

From The National Patient Registry, age, sex and Charlson Comorbidity Index will be retrieved. Mortality during follow-up will be retrieved from The Civil Registration System.

ELIGIBILITY:
Inclusion Criteria:

* Danish adult patient with GERD-diagnosis verified by upper endoscopy 1997-2014

Exclusion Criteria:

* Any diagnosis of cancer in the gastrointestinal tract during follow-up
* Patients with GERD-diagnosis within previous four years or with concomitant diagnosis requiring independent anti-secretory treatment will be excluded (DK25.0-9, DK26.0-9, DK27.0-9, DK22.7 & DE16.4B).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient selection will be done through the Danish National Patient Register. Included will be the period 2000-2015 for a total of 15 years of follow-up.
  All adult Danish patients diagnosed with GERD and GERD-related diagnosis will be identified (ICD-10 DK21.0-21.9B & DK20.9B). Patients with GERD-diagnosis within previous two years or with concomitant diagnosis requiring independent anti-secretory treatment will be excluded (DK25.0-9, DK26.0-9, DK27.0-9, DK22.7 & DE16.4B). To validate GERD-diagnosis, upper endoscopy must have been performed no more than three months before time of diagnosis.
Sampling Method: Probability Sample
Enrollment: 36292 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Treatment of GERD | 2 years after diagnosis
  Medical treatment, surgical treatment or no treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Kolding Hospital, Kolding, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual patient data are by Danish law no allowed to be shared without specific authorization prior to study initiation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT03524781/Prot_SAP_000.pdf